CLINICAL TRIAL: NCT07189546
Title: Development of a Socially Connected Exercise System for Wheelchair Users
Acronym: ParaCycle
Status: Not yet recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: B4249-R
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Exergaming

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — There are no biospecimens collected in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Paracycle Users: Single cohort study. Participants are testing out the Paracycle in their home for 6 weeks.

SUMMARY:
Physical activity (PA) levels among Veterans who use wheelchairs is very low despite the importance of PA in improving overall physical and mental health. Wheelchair users face many barriers to exercise above that of the general population including lack of transportation to PA facilities and programs, social support, motivation and access to accessible fitness equipment and knowledgeable trainers. Home-based fitness products involving access to live and on-demand video instruction and virtual reality applications have become widely popular and beneficial for increasing fitness and motivation among able-bodied individuals during the pandemic however they are not accessible or tailored to the needs of wheelchair users. Therefore, the goal of this project is to develop a home-based upper arm exercise bike that will be compatible with video based instruction and virtual reality real-world riding apps that offer social components and motivational features.

DETAILED DESCRIPTION:
Veterans who use wheelchairs are often prescribed physical activity (PA) in an effort to manage weight and improve cardiovascular health and function however few wheelchair users are currently meeting the recommended amounts of moderate to vigorous aerobic activity (3 times per week ~30 minutes per session). There are many barriers to achieving ample PA including lack of transportation to PA facilities and programs, social support, motivation and access to accessible fitness equipment and knowledgeable trainers. An accessible, motivating, socially supported, and effective exercise option that wheelchair users can participate in from home could help mitigate these barriers to engaging in routine PA. With the onset of the pandemic came a wealth of home-based smart connected exercise devices and fitness apps that enable for interactive video based instruction, virtual/augmented reality world exercise experiences, and integrated social networking features (e.g. group exercise, leaderboards) for the able-bodied market. These applications have been found to improve intrinsic motivation through social support and enjoyment in addition to PA levels and performance. However, these technologies are largely exclusive of persons with disabilities due to the inability to use the connected fitness equipment. Current upper-arm ergometers have limited internet connectivity. Handcycles can be adapted to smart connected bike trainers for use in the home but they require a customized set up that requires a difficult transfer and a lot of space. Therefore, we propose to develop a home-based, smart connected upper-arm ergometer that would enable wheelchairs users to more easily and effectively participate in video and virtual reality-based fitness apps that have social components and motivational features. The specific aims of this study are: 1) to iteratively develop a prototype home-based, smart connected upper-arm cycling trainer (ParaCycle) 2) verify the functionality of the ParaCycle through in lab testing with wheelchair users; and 3) conduct a 6-week in-home pilot study with the refined ParaCycle prototype to evaluate its functionality, safety, utility and device satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* uses a wheelchair
* medically stable (e.g. not currently undergoing rehabilitation or treatment for a medical problem)
* has only the use of their upper limbs for exercise
* lives within one hour driving time from the research center
* has adequate upper limb strength and function to operate an arm ergometer
* has obtained physician clearance to conduct moderate to vigorous exercise
* has room in their home or residence to accommodate the ParaCycle and internet connection

Exclusion Criteria:

* history of fractures or dislocations in the upper extremity from which the participant has not fully recovered
* upper limb pain or injury that interferes with the ability to perform aerobic exercise
* recent hospitalization for any reason (within the past three months)
* history of coronary artery disease, coronary bypass surgery or other cardiorespiratory events or conditions
* likely to experience clinically significant autonomic dysreflexia and/ or orthostatic hypotension in response to exercise
* any other conditions that the persons primary care physician deems is a contraindication to participation in arm ergometry exercise stress testing or moderate to vigorous exercise

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Wheelchair users who have only the use of their arms for exercise
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2027-10-04 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction | After 6 weeks (Trial end)
  Overall reactions to the device on a scale that ranges from 0 (frustrating) to 9 (satisfying).

SECONDARY OUTCOMES:
Adherence Rate | After 6 weeks (Trial end)
  Number of sessions performed during the study period expressed as a percentage of the total number of sessions expected (18).
Retention Rate | After 6 weeks (Trial End)
  Number of participants who complete the study expressed as a percentage of the total number of participants enrolled in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia M Koontz, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data can be made available upon request from the PI and with an approved Data Use Agreement through the VA